CLINICAL TRIAL: NCT05613140
Title: A Pre-post Analysis of Healthcare Resource Utilization and Costs of Care in a New User Cohort of Sacubitril/Valsartan Treated Adult Patients With Chronic Heart Failure
Brief Title: Sacubitril/Valsartan Treated Adult Patients With Chronic Heart Failure
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLCZ696BUS33
Record Dates: First submitted 2022-11-05; First posted 2022-11-14 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Chronic Heart Failure
Keywords: Heart failure,; Medicare Advantage,; Commercial,; HFrEF,; Chronic heart failure
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Cohort 1 - Adult HFrEF patients: adult HFrEF patients who newly initiated sacubitril/valsartan
  Interventions: Drug: sacubitril/valsartan
- Cohort 2 - Adult CHF patients: adult CHF patients who newly initiated sacubitril/valsartan
  Interventions: Drug: sacubitril/valsartan

INTERVENTIONS:
Drug: sacubitril/valsartan — Two study cohorts were constructed to include adult HFrEF patients who newly initiated sacubitril/valsartan (Cohort 1) and adult CHF patients who newly initiated sacubitril/valsartan (Cohort 2).

SUMMARY:
This study evaluated changes in healthcare resource utilization (HCRU) and costs of care within 12 months following initiation of sacubitril/valsartan (sac/val) in commercially insured and Medicare Advantage (MA) lives in the U.S among adult patients with heart failure with reduced ejection fraction (HFrEF) (cohort 1) and adult patients with chronic heart failure (CHF) (cohort 2).

DETAILED DESCRIPTION:
This was a non-interventional, retrospective cohort study using secondary data sources from the Optum Clinformatics® Data Mart (CDM) and 100% files of the CMS Medicare RIFs.

Two study cohorts were constructed to include adult Heart Failure with reduced ejection fraction (HFrEF) patients who newly initiated sacubitril/valsartan (Cohort 1) and adult Chronic Heart Failure (CHF) patients who newly initiated sacubitril/valsartan (Cohort 2).

The date of first prescription fill for sacubitril/valsartan during the cohort identification period was defined as index date. A 12-month washout period was employed to ascertain the "new user" status. The Healthcare Resource Utilization (HCRU) and costs of care outcomes will be measured within both the 12 months post-index period and the 12 months pre-index period.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1 - Adult HFrEF patients

* Newly initiated sacubitril/valsartan during the cohort identification period;
* Presence of an International Classification of Diseases, Tenth revision (ICD-10) diagnosis code for systolic HF (I50.1x, I50.2x, I50.4x) on one inpatient hospital claim or two outpatient medical claims during the cohort identification period;
* That are ≥ 18 years old at index date;
* That are treated with sacubitril/valsartan continuously for a minimum of 90-days following treatment initiation;
* That are continuously enrolled in medical and prescription pharmacy benefits in both the pre-index and post-index period, with any gap in coverage of <45 days allowed.

Cohort 2 - Adult CHF patients

* Newly initiated sacubitril/valsartan during the cohort identification period;
* Presence of ICD-10 diagnosis code for systolic HF or diastolic HF (I50.1x, I50.2x, I50.3x, I50.4x) on one inpatient hospital claim or two outpatient medical claims during the cohort identification period;
* That are ≥ 18 years old at index date;
* That are treated with sacubitril/valsartan continuously for a minimum of 90-days following treatment initiation;
* That are continuously enrolled in medical and prescription pharmacy benefits in both the pre-index and post-index period, with any gap in coverage of <45 days allowed.

Exclusion Criteria:

- Patients who died during the post-index period will be excluded.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with heart failure with reduced ejection fraction (HFrEF) and adult patients with chronic heart failure (CHF)
Sampling Method: Non-Probability Sample
Enrollment: 9230 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
Mean number of Heart Failure - specific hospitalizations of adult HFrEF patients treated with sacubitril/valsartan | Baseline, 12 months post initiation of sacubitril/valsartan
  Number of Heart Failure (HF)-specific hospitalizations was defined as the number of acute inpatient hospitalizations with a primary discharge diagnosis of HF. An acute inpatient hospitalization was defined as a medical claim for an inpatient hospitalization.

SECONDARY OUTCOMES:
Mean number of HF - related hospitalizations of adult HFrEF patients treated with sacubitril/valsartan | Baseline, 12 months post initiation of sacubitril/valsartan
  Number of HF-related hospitalizations was defined as the number of acute inpatient hospitalizations with a discharge diagnosis of HF in any position.
Mean number of all-cause hospitalizations of adult HFrEF patients treated with sacubitril/valsartan | Baseline, 12 months post initiation of sacubitril/valsartan
  Number of all-cause hospitalizations was as the number of acute inpatient hospitalizations for any reason.
Mean number of Urgent Heart Failure (UHF) visits of adult HFrEF patients treated with sacubitril/valsartan | Baseline, 12 months post initiation of sacubitril/valsartan
  An UHF visit was defined as any of the following:
  i) a patient with a place of service (POS) code 20, which corresponds to urgent care facility ii) a patient with an ER visit that was outpatient (POS code = 22, 23), identified from revenue codes: 0450, 0451, 0452, 0456 or 0459 iii) a patient with an urgent care clinic visit that was outpatient (POS code = 22, 23), identified from revenue codes: 0516 or 0526 iv) a patient with a hospital observational stay (POS code = 22, 23), identified from revenue code 0762
Mean number of Worsening Heart Failure (WHF) episodes of adult HFrEF patients treated with sacubitril/valsartan | Baseline, 12 months post initiation of sacubitril/valsartan
  Number of WHF episodes was defined as a composite outcome of HF-specific hospitalizations and UHF visits.
Mean costs of HF-specific hospitalizations of adult HFrEF patients treated with sacubitril/valsartan | Baseline, 12 months post initiation of sacubitril/valsartan
  Costs of HF-specific hospitalizations was defined as the sum of payer paid amounts for acute inpatient hospitalizations with a primary discharge diagnosis of HF.
Mean costs of HF-related hospitalizations of adult HFrEF patients treated with sacubitril/valsartan | Baseline, 12 months post initiation of sacubitril/valsartan
  Costs of HF-related hospitalizations were defined as the sum of payer paid amounts for acute inpatient hospitalizations with a discharge diagnosis of HF in any position.
Mean costs of all-cause hospitalizations of adult HFrEF patients treated with sacubitril/valsartan | Baseline, 12 months post initiation of sacubitril/valsartan
  Costs of all-cause hospitalizations were defined as the sum of payer paid amounts for acute inpatient hospitalizations for any reason.
Mean costs of UHF visits of adult HFrEF patients treated with sacubitril/valsartan | Baseline, 12 months post initiation of sacubitril/valsartan
  Costs of UHF visits were defined as the sum of payer paid amounts for UHF visits.
Mean costs of WHF episodes of adult HFrEF patients treated with sacubitril/valsartan | Baseline, 12 months post initiation of sacubitril/valsartan
  Costs of WHF episodes were defined as the sum of payer paid amounts for HF-specific hospitalizations and UHF visits.
Mean HF-specific costs of adult HFrEF patients treated with sacubitril/valsartan | Baseline, 12 months post initiation of sacubitril/valsartan
  HF-related costs were defined as the sum of payer paid amounts for medical claims with a diagnosis of HF in any position.
Mean all-cause medical costs of adult HFrEF patients treated with sacubitril/valsartan | Baseline, 12 months post initiation of sacubitril/valsartan
  All-cause medical costs were defined as the sum of payer paid amounts for all medical claims.
Mean all-cause pharmacy costs of adult HFrEF patients treated with sacubitril/valsartan | Baseline, 12 months post initiation of sacubitril/valsartan
  All-cause pharmacy costs were defined as the sum of payer paid amounts for all pharmacy claims.
Mean all-cause total cost of care of adult HFrEF patients treated with sacubitril/valsartan | Baseline, 12 months post initiation of sacubitril/valsartan
  All-cause total cost of care were defined as the sum of all-cause medical costs and all-cause pharmacy costs.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CLCZ696BUS33 from the Novartis Clinical Trials Website — http://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17992